CLINICAL TRIAL: NCT06800131
Title: A Phase I, Randomized, Open-Label, Active-Control Study to Evaluate Safety, Tolerability, and Immunogenicity of Recombinant Hepatitis B Vaccine Delivered Trans-dermally by Microneedle Array Patch (MAP) in Healthy Adults
Brief Title: Hepatitis B Vaccine Delivered Trans-dermally by MAP
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: QuadMedicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVI QMHepB-01
Record Dates: First submitted 2025-01-02; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis B Vaccine
Keywords: Microneedle array patch
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: Healthy adults between 19 to 40 years of age will be screened for eligibility criteria. A total of 40 subjects will be enrolled, 30 subjects administered trans-dermally via MAP and 10 subjects administered with active comparator vaccine via intramuscular injection. Subjects will be randomized to either transdermal MAP arm or IM Injection arm with ratio of 3:1. At Day 0, subject will receive 1st vaccination, followed by 2nd and 3rd injection at W4 and W26, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine administered trans-dermally via MAP (Experimental): Manufacturer: QuadMedicine Inc. Form: Microarray needle patch Appearance: Patch Dose: one patch contains 20μg of HbsAg (drug substance manufactured by LG Chemical)
  Route: Intra-dermal (Skin application)Each patch of vaccine contains the following components:
  * HBsAg 20μg (drug substance manufactured by LG Chemical)
  * Sodium carboxymethyl cellulose (CMC Na): 20μg
  * Trehalose: 400μg
  Interventions: Device: Hepatitis B Vaccine administered trans-dermally via Microneedle Array Patch (MAP)
- Active comparator vaccine via intramuscular injection (Active Comparator): Euvax B™ (LG Chemical) is a white, slightly opalescent suspension.1 ml of the above vaccine contains:
  * Active ingredient: Purified HBsAg 20µg
  * Adjuvant: Aluminum Hydroxide Gel 0.5 mg
  * Excipients: Potassium phosphate, Sodium phosphate, Sodium chloride
  Interventions: Biological: Active comparator vaccine via intramuscular injection

INTERVENTIONS:
Device: Hepatitis B Vaccine administered trans-dermally via Microneedle Array Patch (MAP) — A total of 40 subjects will be enrolled, 30 subjects administered trans-dermally via Microneedle Array Patch (MAP).
  Arms: Vaccine administered trans-dermally via MAP
Biological: Active comparator vaccine via intramuscular injection — 10 subjects administered with active comparator vaccine via intramuscular injection.
  Arms: Active comparator vaccine via intramuscular injection

SUMMARY:
This is Phase I, randomized, open-label, active-controlled study to evaluate the safety, tolerability, and immunogenicity of a hepatitis B vaccine administered trans-dermally via microneedle array patch (MAP) compared to the intra-muscular (IM) hepatitis B vaccine (Euvax B™), administered at Day (D) 0, Week (W) 4, W26 among healthy adults aged 19 to 40 years in the Republic of Korea.

DETAILED DESCRIPTION:
This is Phase I, randomized, open-label, active-controlled study to evaluate the safety, tolerability, and immunogenicity of a hepatitis B vaccine administered trans-dermally via microneedle array patch (MAP) compared to the intra-muscular (IM) hepatitis B vaccine (Euvax B™), administered at Day (D) 0, Week (W) 4, W26 among healthy adults aged 19 to 40 years in the Republic of Korea.

Healthy adults between 19 to 40 years of age will be screened for eligibility criteria. A total of 40 subjects will be enrolled, 30 subjects administered trans-dermally via MAP and 10 subjects administered with active comparator vaccine via intramuscular injection. Subjects will be randomized to either transdermal MAP arm or IM Injection arm with ratio of 3:1. At D0, subject will receive 1st vaccination, followed by 2nd and 3rd vaccination at W4 and W26, respectively.

For the first five (5) subjects who completed Week 1 visit, all available clinical laboratory and adverse event data will be reviewed in a rolling manner by Study Medical Monitor and Site PI. Further enrollment will be paused during safety review by the independent data safety monitoring board (DSMB). If there are no safety findings judged to be of clinical concern and has not met the trial halting criteria specified in the protocol section 10.1.4, subsequent dosing (2nd dose) will be opened for the first 5 subjects and enrollment of the remaining 35 subjects will begin. If any of the halting rules are met, the study will be halted immediately for DSMB review/recommendation.

After all enrolled subjects complete Visit 6 (4 weeks after 3rd dose), the DSMB will be convened to review the safety and immunogenicity data once available to look at the sero-protection rates and titers to formulate further recommendations and be diligent in case there are non-responders to MAP Hep B vaccine. All SMC and DSMB meetings will be conducted per SMC and DSMB charter, respectively.

The solicited and unsolicited adverse events will be recorded up to 7 days and 28 days, respectively for each injection. Relatedness of all adverse events that occurred in the MAP arm will be assessed to biologics component (active ingredient; HBsAg) as well as medical device component (microneedle patch). Serious adverse events (SAEs) and adverse events of special interest (AESIs) will be collected throughout the study.

Should the criteria for any temporary pause of immunization rule be met, at any time, further enrollment and administration of investigational product will be paused for further evaluation. The Sponsor will consult the DSMB, if needed, to determine whether to enroll and/or continue enrollment and/or dosing of remainder of the subjects.

All subjects will be followed for 52 weeks following the 1st vaccination. Week 52 of the last subject enrolled will be the End of Study (EOS) visit.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate with investigator, and to provide informed consent and have signed Informed Consent Form (ICF) prior to screening procedures
2. Adults aged 19 to 40 years
3. Judged to be healthy by the Investigator on the basis of medical history, physical examination, screening laboratory results and vital signs performed at screening visit
4. Able and willing to comply with all study procedures during the study period
5. Negative serological tests for Hepatitis B surface antigen (HBsAg), Hepatitis B surface antibody (Anti-HBs), antibody to Hepatitis B core antibody (anti-HBc), Hepatitis C antibody and Human Immunodeficiency Virus (HIV) antibody at screening

Exclusion Criteria:

1. Pregnant or breastfeeding, or intending to become pregnant or father children within the projected duration of the trial starting with the screening visit until 3 months following last dose
2. Positive serum pregnancy test at screening or positive urine pregnancy test prior at dosing visit
3. Self-reported history of Hepatitis B vaccination beyond childhood Hepatitis B immunization series
4. Currently participating in or has participated in a study with an investigational product administered within 6 months preceding Day 0
5. Body mass index (BMI) <18 or >30 kg/m²
6. Current or history of the following medical conditions:

   * Diagnosis of malignancy within 5 years of screening
   * Diagnosis of diabetes mellitus or HbA1c ≥7%
   * Liver transaminases > 2 times the upper limit of the normal range
   * Impaired renal function as creatinine >120 mmol/L or calculated glomerular filtration rate <60mls/min
   * Use of immunoglobulin or blood products in last 3 months
   * History of severe allergic reaction or anaphylaxis after immunization or administration of any medical products that contain drug substances of investigational product

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2026-08-05 (Estimated); Study Completion 2026-11-05 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of investigational product (QMV-24KRP) | Within 52 weeks of the first IP administration
  * Occurrence of any SAEs from the time of the first vaccination through the final visit
  * Occurrence of immediate reaction (reactogenicity event) within 30 minutes post each vaccination.
  * Occurrence of solicited local and systemic reactions within 7 days post each vaccination
  * Occurrence of unsolicited AEs within 28 days post each vaccination

SECONDARY OUTCOMES:
To assess anti-HBs response before the first vaccination and after each injection of QMV-24KRP | Within 52 weeks of the first IP administration
  * Percentage of subjects achieving sero-protection level (defined as anti-HBs antibody titer ≥ 10 IU/L) at Week 30 (4 weeks post third-dose vaccination)
  * Percentage of subjects achieving sero-protection level (defined as anti-HBs antibody titer ≥10 IU/L) at Week 52 (26 weeks post third-dose vaccination)
  * Percentage of subjects considered as good responder (defined as anti-HBs ≥ 100 IU/L) at Week 30 or Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Hee Soo Kim, Principal Investigator — Non-governmental Organization

IPD SHARING:
Plan to Share IPD: No